CLINICAL TRIAL: NCT06743217
Title: IS THERE A DIFFERENCE IN TEXTBOOK OUTCOMES OF EMERGENCY CHOLECYSTECTOMY IN ELDERLY PATIENTS COMPARED TO OTHERS
Brief Title: TEXTBOOK OUTCOMES OF EMERGENCY CHOLECYSTECTOMIES IN ELDERLY PATIENTS
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasir Musa Kesgin, MD, MD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2024-165
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Acute Cholecystitis
Keywords: Acute Cholecystitis; Textbook Outcome; Emergency Surgery
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: All patients which are younger than 65 years old and underwent emergency cholecystectomy between 2020 and 2024
- Group B- Elderly Group: All patients ≥ 65 years old and underwent emergency cholecystectomy between 2020 and 2024

SUMMARY:
Textbook outcome is a measure used to assess the quality of surgical practice. The goal of this observational study is to compare textbook outcomes of elderly patients (≥65 years) in emergency cholecystectomies with younger patients(<65 years ) via using aforementioned criteria

DETAILED DESCRIPTION:
Textbook outcome is a measure used to assess the quality of surgical practice and has been implemented in various areas of surgical literature. It is defined as an uneventful operative and postoperative period that leads to successful surgery without negative outcomes. There is still no consensus on the textbook outcome concept for emergency cholecystectomy. SPRIMACC Collaborative Study has presented and offered a list of textbook outcome criteria.

Their proposal was: no 30-day mortality, no 30-day postoperative complications (any CD≥I is considered non-TO), no readmission within 30 days, and hospital stay≤7 days (75th percentile) and full laparoscopic surgery.

The goal of this observational study is to compare textbook outcomes of elderly patients (≥65 years) in emergency cholecystectomies with younger patients(<65 years ) via using aforementioned criteria

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent emergency cholecystectomy with a diagnosis of acute choleystitis

Exclusion Criteria:

* Patients underwent open surgery directly. Patients diagnosed as malignant postoperatively in the pathology report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old and underwent emergency cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Textbook Outcome | 30 days
  The Textbook Outcome criteria for emergency cholecystectomy in this study were patients have these criteria: no 30-day mortality, no 30-day postoperative complications, no readmission within 30 days, hospital stay≤7 days and full laparoscopic surgery

SECONDARY OUTCOMES:
Subtotal cholecystectomy | 1 day
  Patients underwent emergency surgery with a diagnosis of acute cholecystitis and subtotal cholecystectoym performed
Postoperative Serious Complications | 30 days
  Postoperative complications that have a Clavien-Dindo Score ≥3 were accepted as serious complication.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Musa Kesgin, MD, Study Chair — University of Health Sciences, Kanuni Sultan Suleyman Training and Research Hospital, Department of General Surgery, Istanbul,Türkiye
Locations (1):
- University of Health Sciences, Kanuni Sultan Suleyman Training and Research Hospital, Department of General Surgery, Istanbul, Turkey (Türkiye)